CLINICAL TRIAL: NCT00405704
Title: Randomized Intervention for Children With Vesicoureteral Reflux (RIVUR)
Acronym: RIVUR
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: National Institute of Diabetes and Digestive and Kidney Diseases (NIDDK) (NIH)
Collaborators: University of North Carolina, Chapel Hill (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: DK074059 (IND); U01DK074059 (NIH)
Record Dates: First submitted 2006-11-29; First posted 2006-11-30 (Estimated); Results first posted 2015-04-16 (Estimated); Last update posted 2020-04-21 (Actual); Status verified 2020-04

CONDITIONS: Vesicoureteral Reflux; Urinary Tract Infections
Keywords: Vesicoureteral Reflux; Urinary Tract Infections; Renal Scarring; Antibiotic Resistance; Controlled Clinical Trial; Trimethoprim-Sulfamethoxazole; Children
MeSH Terms: conditions — Vesico-Ureteral Reflux; Urinary Tract Infections | interventions — Trimethoprim, Sulfamethoxazole Drug Combination

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Trimethoprim-Sulfamethoxazole (Active Comparator): Cherry-flavored liquid suspension with 3 mg of trimethoprim plus 15 mg sulfamethoxazole per kilogram of body weight, taken once daily.
  Interventions: Drug: Trimethoprim-Sulfamethoxazole
- Placebo (Placebo Comparator): Cherry-flavored liquid suspension matched to active comparator.
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Trimethoprim-Sulfamethoxazole — Cherry-flavored liquid suspension with 3 mg of trimethoprim plus 15 mg sulfamethoxazole per kilogram of body weight, taken once daily.
  Other Names: Sulfatrim; Bactrim
  Arms: Trimethoprim-Sulfamethoxazole
Drug: Placebo — Cherry flavored liquid suspension matched to active comparator.
  Arms: Placebo

SUMMARY:
In this 2-year, multisite, randomized, placebo-controlled trial involving 607 children with vesicoureteral reflux that was diagnosed after a first or second febrile or symptomatic urinary tract infecton, we evaluated the efficacy of Trimethoprim-Sulfamethoxazole (TMP-SMZ) prophylaxis in preventing recurrences (primary outcome). Secondary outcomes were renal scarring, treatment failure (a composite of recurrences and scarring), and antimicrobial resistance.

DETAILED DESCRIPTION:
This multicenter, randomized, double-blind, placebo-controlled trial was designed to determine whether daily antimicrobial prophylaxis is superior to placebo in preventing recurrence of urinary tract infection (UTI) in children with vesicoureteral reflux (VUR). Eligibility criteria are described elsewhere. Patients were randomly assigned to treatment for 2 years with daily antimicrobial prophylaxis (trimethoprim-sulfamethoxazole) or placebo. The study was designed to recruit 600 children (approximately 300 in each treatment group). The protocol encouraged prompt evaluation of children with UTI symptoms and early therapy of culture-proven UTIs. It was expected that approximately 10% of children will have to discontinue study medication due to allergic reactions. Assuming a 20% placebo event rate and 10% non-compliance rate, the study has 83% power to detect an absolute 10% event rate in the antimicrobial prophylaxis group. If the placebo event rate is instead 25%, power is 97% to detect an absolute 10% event rate in the treated group, even if non-compliance is as high as 15%. The primary analysis is intention-to-treat with missing outcome data analyzed as UTI.

In addition to collecting follow-up data on urinary tract infections, renal scarring and antimicrobial resistance, quality of life, compliance, safety parameters, utilization of health resources, and change in VUR were assessed periodically throughout the study.

ELIGIBILITY:
Inclusion Criteria:

* Age at randomization: at least 2 months, but less than 6 years of age. Note that children as young as 1 month were screened for the study.
* Diagnosed first or second febrile or symptomatic UTI within 112 days prior to randomization
* Presence of Grade I- IV VUR based on radiographic voiding cystourethrogram (VCUG) performed within 112 days of diagnosis of index UTI.
* Appropriately treated index febrile or symptomatic UTI

Exclusion Criteria:

* Index UTI diagnosis more than 112 days prior to randomization
* History of more than two UTIs prior to randomization
* For patients less than 6 months of age at randomization, gestational age less than 34 weeks
* Co-morbid urologic anomalies
* Hydronephrosis, SFU Grade 4
* Ureterocele
* Urethral valve
* Solitary kidney
* Profoundly decreased renal size unilaterally on ultrasound (based on 2 standard deviations below the mean for age and length) performed within 112 days after diagnosis of index UTI
* Multicystic dysplastic kidney
* Neurogenic bladder
* Pelvic kidney or fused kidney
* Known sulfa allergy, inadequate renal or hepatic function, Glucose-6-phosphate dehydrogenase deficiency or other conditions that are contraindications for use of TMP-SMZ
* History of other renal injury/disease
* Unable to complete the study protocol
* Congenital or acquired immunodeficiency
* Underlying anomalies or chronic diseases that could potentially interfere with response to therapy such as chronic gastrointestinal conditions (i.e., malabsorption, inflammatory bowel disease), liver or kidney failure, or malignancy.
* Complex cardiac disease as defined in the Manual of Procedures.
* Any known syndromes associated with VUR or bladder dysfunction
* Index UTI not successfully treated
* Unlikely to complete follow-up
* Family history of anaphylactic reaction to sulfa medications

Ages: 2 Months to 71 Months | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 607 (Actual)
Dates: Start 2007-05 (Actual); Primary Completion 2013-06 (Actual); Study Completion 2014-05 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Sahar Fathallah, MD, Principal Investigator — University of Alabama, Birmingham, AL; Myra A Carpenter, PhD, Principal Investigator — University of NC at Chapel Hill, Chapel Hill, NC; Caleb P. Nelson, MD, MPH, Principal Investigator — Children's Hospital of Boston, Boston, MA; Eileen Brewer, MD, Principal Investigator — Texas Children's Hospital, Houston, TX; Saul P Greenfield, MD, Principal Investigator — Women and Children's Hospital of Buffalo, Buffalo, NY; Alejandro Hoberman, MD, Principal Investigator — Children's Hospital of Pittsburgh, Pittsburgh, PA; Ron Keren, MD, MPH, Principal Investigator — Children's Hospital of Philadelphia, Philadelphia, PA; Bradley P Kropp, MD, Principal Investigator — University of Oklahoma, Oklahoma City, OK; Ranjiv Mathews, MD, Principal Investigator — Johns Hopkins University; Tej K Mattoo, MD,DCH, FRCP, Principal Investigator — Wayne State University School of Medicine, Detroit, MI; H. Gil Rushton, MD, FAAP, Principal Investigator — Children's National Research Institute; Mary Ann Queen, MD, Principal Investigator — Children's Mercy Hospital Kansas City; Russell W Chesney, MD, Study Chair — Le Bonheur Children's Medical Center, Memphis, TN; Steven J Skoog, MD FACS,FAAP, Principal Investigator — Oregon Health & Science University, Portland, OR; Amy Renwick, MD, Principal Investigator — Alfred I. duPont Hospital for Children, Wilmington, DE; Earl Y. Cheng, MD, Principal Investigator — Ann & Robert H. Lurie Children's Hospital of Chicago, Chicago, IL; Milan Nadkarni, MD, Principal Investigator — Wake Forest University Baptist Medical Center, Winston-Salem, NC; Caleb P Nelson, MD, MPH, Principal Investigator — Children's Hospital of Boston, Boston, MA; William R DeFoor, Jr, MD, MPH, Principal Investigator — Cincinnati Children's Hospital, Cincinnati, OH; Dan McMahon, MD, Principal Investigator — Akron Children's Hospital, Akron, OH; Ross Decter, MD, Principal Investigator — Penn State Hershey Medical Center, Hershey, PA; Sharon M Bartosh, MD, Principal Investigator — University of Wisconsin, Madison
Locations (19):
- United States (19):
  - University of Alabama, Birmingham, Alabama
  - Alfred I. duPont Hospital for Children, Wilmington, Delaware
  - Children's National Medical Center, Washington D.C., District of Columbia
  - Ann & Robert Lurie Children's Hospital of Chicago, Chicago, Illinois
  - Johns Hopkins School of Medicine, Baltimore, Maryland
  - Children's Hospital of Boston, Boston, Massachusetts
  - Children's Hospital of Michigan, Detroit, Michigan
  - Children's Mercy Hospital, Kansas City, Missouri
  - Women and Children's Hospital of Buffalo, Buffalo, New York
  - Wake Forest University Baptist Medical Center, Winston-Salem, North Carolina
  - Akron Children's Hospital, Akron, Ohio
  - Cincinnati Children's Hospital, Cincinnati, Ohio
  - University of Oklahoma, Oklahoma City, Oklahoma
  - Oregon Health & Science University, Portland, Oregon
  - Penn State Hershey Medical Center, Hershey, Pennsylvania
  - Children's Hospital of Philadelphia, Philadelphia, Pennsylvania
  - Children's Hospital of Pittsburgh, Pittsburgh, Pennsylvania
  - Texas Children's Hospital, Houston, Texas
  - University of Wisconsin Children's Hospital, Madison, Wisconsin

IPD SHARING:
Plan to Share IPD: Yes
Data are available at the NIDDK Central Repository: https://repository.niddk.nih.gov/studies/rivur/?query=rivur
URL: https://repository.niddk.nih.gov/studies/rivur/?query=rivur

REFERENCES:
- [Background] Ziessman HA, Majd M. Importance of methodology on (99m)technetium dimercapto-succinic acid scintigraphic image quality: imaging pilot study for RIVUR (Randomized Intervention for Children With Vesicoureteral Reflux) multicenter investigation. J Urol. 2009 Jul;182(1):272-9. doi: 10.1016/j.juro.2009.02.144. Epub 2009 May 17. PMID 19450818
- [Background] Mathews R, Carpenter M, Chesney R, Hoberman A, Keren R, Mattoo T, Moxey-Mims M, Nyberg L, Greenfield S. Controversies in the management of vesicoureteral reflux: the rationale for the RIVUR study. J Pediatr Urol. 2009 Oct;5(5):336-41. doi: 10.1016/j.jpurol.2009.05.010. Epub 2009 Jul 1. PMID 19570724
- [Background] Keren R, Carpenter MA, Hoberman A, Shaikh N, Matoo TK, Chesney RW, Matthews R, Gerson AC, Greenfield SP, Fivush B, McLurie GA, Rushton HG, Canning D, Nelson CP, Greenbaum L, Bukowski T, Primack W, Sutherland R, Hosking J, Stewart D, Elder J, Moxey-Mims M, Nyberg L. Rationale and design issues of the Randomized Intervention for Children With Vesicoureteral Reflux (RIVUR) study. Pediatrics. 2008 Dec;122 Suppl 5(Suppl 5):S240-50. doi: 10.1542/peds.2008-1285d. PMID 19018048
- [Background] Greenfield SP, Chesney RW, Carpenter M, Moxey-Mims M, Nyberg L, Hoberman A, Keren R, Matthews R, Mattoo T. Vesicoureteral reflux: the RIVUR study and the way forward. J Urol. 2008 Feb;179(2):405-7. doi: 10.1016/j.juro.2007.10.100. No abstract available. PMID 18076937
- [Background] Chesney RW, Carpenter MA, Moxey-Mims M, Nyberg L, Greenfield SP, Hoberman A, Keren R, Matthews R, Matoo TK; members of the RIVUR Steering Committee. Randomized Intervention for Children With Vesicoureteral Reflux (RIVUR): background commentary of RIVUR investigators. Pediatrics. 2008 Dec;122 Suppl 5(0 5):S233-9. doi: 10.1542/peds.2008-1285c. PMID 19018047
- [Background] Keren R. Pediatrics. RIVUR trial. Introduction. Pediatrics. 2008 Dec;122 Suppl 5:S231-2. doi: 10.1542/peds.2008-1285b. No abstract available. PMID 19086141
- [Background] Greenfield SP, Carpenter MA, Chesney RW, Zerin JM, Chow J. The RIVUR voiding cystourethrogram pilot study: experience with radiologic reading concordance. J Urol. 2012 Oct;188(4 Suppl):1608-12. doi: 10.1016/j.juro.2012.06.032. Epub 2012 Aug 19. PMID 22910235
- [Background] Hoberman A, Shaikh N, Bhatnagar S, Haralam MA, Kearney DH, Colborn DK, Kienholz ML, Wang L, Bunker CH, Keren R, Carpenter MA, Greenfield SP, Pohl HG, Mathews R, Moxey-Mims M, Chesney RW. Factors that influence parental decisions to participate in clinical research: consenters vs nonconsenters. JAMA Pediatr. 2013 Jun;167(6):561-6. doi: 10.1001/jamapediatrics.2013.1050. PMID 23546617
- [Background] Bhatnagar S, Hoberman A, Kearney DH, Shaikh N, Moxey-Mims MM, Chesney RW, Carpenter MA, Greenfield SP, Keren R, Mattoo TK, Mathews R, Gravens-Mueller L, Ivanova A. Development and impact of an intervention to boost recruitment in a multicenter pediatric randomized clinical trial. Clin Pediatr (Phila). 2014 Feb;53(2):151-7. doi: 10.1177/0009922813506961. Epub 2013 Oct 22. PMID 24151147
- [Background] Chesney RW, Patters AB. Childhood vesicoureteral reflux studies: registries and repositories sources and nosology. J Pediatr Urol. 2013 Dec;9(6 Pt A):731-7. doi: 10.1016/j.jpurol.2012.09.003. Epub 2012 Oct 5. PMID 23044377
- [Result] Carpenter MA, Hoberman A, Mattoo TK, Mathews R, Keren R, Chesney RW, Moxey-Mims M, Greenfield SP; RIVUR Trial Investigators. The RIVUR trial: profile and baseline clinical associations of children with vesicoureteral reflux. Pediatrics. 2013 Jul;132(1):e34-45. doi: 10.1542/peds.2012-2301. Epub 2013 Jun 10. PMID 23753091
- [Result] RIVUR Trial Investigators; Hoberman A, Greenfield SP, Mattoo TK, Keren R, Mathews R, Pohl HG, Kropp BP, Skoog SJ, Nelson CP, Moxey-Mims M, Chesney RW, Carpenter MA. Antimicrobial prophylaxis for children with vesicoureteral reflux. N Engl J Med. 2014 Jun 19;370(25):2367-76. doi: 10.1056/NEJMoa1401811. Epub 2014 May 4. PMID 24795142
- [Derived] Primack W, Bukowski T, Sutherland R, Gravens-Mueller L, Carpenter M. What Urinary Colony Count Indicates a Urinary Tract Infection in Children? J Pediatr. 2017 Dec;191:259-261.e1. doi: 10.1016/j.jpeds.2017.08.012. Epub 2017 Sep 28. PMID 28967387
- [Derived] Keren R, Shaikh N, Pohl H, Gravens-Mueller L, Ivanova A, Zaoutis L, Patel M, deBerardinis R, Parker A, Bhatnagar S, Haralam MA, Pope M, Kearney D, Sprague B, Barrera R, Viteri B, Egigueron M, Shah N, Hoberman A. Risk Factors for Recurrent Urinary Tract Infection and Renal Scarring. Pediatrics. 2015 Jul;136(1):e13-21. doi: 10.1542/peds.2015-0409. Epub 2015 Jun 8. PMID 26055855
- See also: RIVUR trial web site — http://www.rivur.net

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Trimethoprim-Sulfamethoxazole | Placebo
Started | 302 | 305
Completed Outcome Renal Scan | 227 | 235
Completed Assessments for New Scarring | 220 | 227
Outcome Stool Assessed | 203 | 210
Recurrent UTI With E. Coli | 30 | 57
Recurrent UTI With TMP-SMZ Panel | 38 | 69
Completed | 261 | 259
Not Completed | 41 | 46

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Trimethoprim-Sulfamethoxazole | Placebo | Total
Number analyzed (Participants) | 302 | 305 | 607
Age, Continuous [Median (Inter-Quartile Range); unit: months] | 12 [5 to 31] | 12 [6 to 30] | 12 [6 to 31]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 277 | 281 | 558
  Male | 25 | 24 | 49
Region of Enrollment [Number; unit: participants]
  United States | 302 | 305 | 607

OUTCOME MEASURES:

1. Primary Outcome: Recurrent Febrile or Symptomatic Urinary Tract Infection During 2-year Follow-up
Time Frame: 2 years
Measure: Number; unit: participants
Arm/Group | Trimethoprim-Sulfamethoxazole | Placebo
Number analyzed (Participants) | 302 | 305
participants | 39 | 72
Statistical Analysis 1: Comparison: Trimethoprim-Sulfamethoxazole vs Placebo; Test type: Superiority or Other; p < 0.001, Log Rank

2. Secondary Outcome: Outcome Renal Scarring
Description: Renal scarring was defined as a decreased uptake of tracer that was associated with loss of contours or the presence of cortical thinning. Outcome dimercaptosuccinic acid (DMSA) scan was performed at 2 years after enrollment or 3-4 months after the child had met treatment failure criteria.
Time Frame: 2 years
Population: The analysis population excluded 75 subjects in the trimethoprim-sulfamethoxazole group and 70 subjects in the placebo group who did not have an outcome dimercaptosuccinic acid scan.
Measure: Number; unit: participants
Arm/Group | Trimethoprim-Sulfamethoxazole | Placebo
Number analyzed (Participants) | 227 | 235
participants | 27 | 24
Statistical Analysis 1: Comparison: Trimethoprim-Sulfamethoxazole vs Placebo; Test type: Superiority or Other; p = 0.55, Cochran-Mantel-Haenszel

3. Secondary Outcome: Severe Renal Scarring on Outcome Scan
Description: Severe renal scarring was defined as scarring in more than 4 of 12 segments in at least one kidney or global atrophy characterized by diffusely scarred and shrunken kidney. Outcome DMSA scan performed at 2 years after enrollment or 3-4 months after the child had met treatment failure criteria.
Time Frame: 2 years
Population: as for outcome 2
Measure: Number; unit: participants
Arm/Group | Trimethoprim-Sulfamethoxazole | Placebo
Number analyzed (Participants) | 227 | 235
participants | 9 | 6
Statistical Analysis 1: Comparison: Trimethoprim-Sulfamethoxazole vs Placebo; Test type: Superiority or Other; p = 0.37, Cochran-Mantel-Haenszel

4. Secondary Outcome: New Renal Scarring on Outcome Scan
Description: New renal scarring was defined as scarring on the outcome renal scan with technetium -99m-labeled dimercaptosuccinic acid that was not present at baseline. Outcome DMSA scan performed at 2 years after enrollment or 3-4 months after the child had met treatment failure criteria.
Time Frame: 2 years
Population: The analysis population excluded 82 subjects in the trimethoprim-sulfamethoxazole group and 78 subjects in the placebo group who did not have an outcome dimercaptosuccinic acid scan.
Measure: Number; unit: participants
Arm/Group | Trimethoprim-Sulfamethoxazole | Placebo
Number analyzed (Participants) | 220 | 227
participants | 18 | 19
Statistical Analysis 1: Comparison: Trimethoprim-Sulfamethoxazole vs Placebo; Test type: Superiority or Other; p = 0.94, Cochran-Mantel-Haenszel

5. Secondary Outcome: Treatment Failure Composite
Description: Treatment failure was defined as the occurrence of two febrile urinary tract infections (UTIs), one febrile UTI and three symptomatic UTIs, four symptomatic UTIs, or new or worsening renal scarring on an interim scan (e.g,, the 12-month visit); renal scans from the 2-year visit are NOT considered in the treatment failure criteria.
Time Frame: 2 years
Measure: Number; unit: participants
Arm/Group | Trimethoprim-Sulfamethoxazole | Placebo
Number analyzed (Participants) | 302 | 305
participants | 14 | 27
Statistical Analysis 1: Comparison: Trimethoprim-Sulfamethoxazole vs Placebo; Test type: Superiority or Other; p = 0.04, Log Rank

6. Secondary Outcome: Presence of E.Coli Resistant to Trimethoprim-Sulfamethoxazole (TMP-SMZ) (Based on Rectal Swab)
Time Frame: 2 years
Population: The analysis population excluded 99 subjects in the trimethoprim-sulfamethoxazole group and 95 subjects in the placebo group who did not have stool analyzed at the outcome visit.
Measure: Number; unit: participants
Arm/Group | Trimethoprim-Sulfamethoxazole | Placebo
Number analyzed (Participants) | 203 | 210
participants | 56 | 41
Statistical Analysis 1: Comparison: Trimethoprim-Sulfamethoxazole vs Placebo; Test type: Superiority or Other; p = 0.065, Cochran-Mantel-Haenszel

7. Secondary Outcome: Recurrent Febrile or Symptomatic UTI With Resistant E. Coli
Time Frame: 2 years
Population: The analysis population is restricted to the 30 subjects in the trimethoprim-sulfamethoxazole (TMP-SMZ) group and 57 subjects in the placebo group who had a recurrent UTI with E. coli for which sensitivity to TMP-SMZ was assessed.
Measure: Number; unit: participants
Arm/Group | Trimethoprim-Sulfamethoxazole | Placebo
Number analyzed (Participants) | 30 | 57
participants | 19 | 11
Statistical Analysis 1: Comparison: Trimethoprim-Sulfamethoxazole vs Placebo; Test type: Superiority or Other; p < 0.001, Cochran-Mantel-Haenszel

8. Secondary Outcome: Recurrent Febrile or Symptomatic UTI With Any Resistant Pathogen
Time Frame: 2 years
Population: The analysis population is restricted to the 38 subjects in the trimethoprim-sulfamethoxazole (TMP-SMZ) group and 69 subjects in the placebo group who had a recurrent UTI with an organism for which sensitivity to TMP-SMZ was assessed.
Measure: Number; unit: participants
Arm/Group | Trimethoprim-Sulfamethoxazole | Placebo
Number analyzed (Participants) | 38 | 69
participants | 26 | 17
Statistical Analysis 1: Comparison: Trimethoprim-Sulfamethoxazole vs Placebo; Test type: Superiority or Other; p < 0.001, Cochran-Mantel-Haenszel

ADVERSE EVENTS:
Time Frame: 2 years
Arm/Group | Trimethoprim-Sulfamethoxazole | Placebo
Serious Adverse Events (participants affected / at risk) | 0/302 | 0/305
Other Adverse Events (participants affected / at risk) | 79/302 | 105/305
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Trimethoprim-Sulfamethoxazole (N=302) | Placebo (N=305)
Fever (General disorders) | 43 (58) | 55 (80)
Otitis Media (General disorders) | 13 (18) | 24 (33)
Pharyngitis (General disorders) | 19 (25) | 14 (20)
Rash (General disorders) | 23 (30) | 23 (26)
Viral Infection (General disorders) | 14 (14) | 16 (20)
Diarrhea (General disorders) | 11 (14) | 19 (27)

LIMITATIONS AND CAVEATS:
Results may not apply to children with different demographic or clinical characteristics or in locales where choice of TMP-SMZ may be limited by susceptibility patterns or clinical acceptability. Some subgroup analyses had limited statistical power.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No